CLINICAL TRIAL: NCT00067912
Title: Duloxetine Versus Venlafaxine Extended Release in the Treatment of Major Depressive Disorder
Brief Title: Duloxetine vs. Active Comparator for the Treatment of Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7999; F1J-MC-HMCQ
Record Dates: First submitted 2003-08-29; First posted 2003-09-03 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride
Drug: Venlafaxine Extended Release

SUMMARY:
How duloxetine compares to a medication currently available for the treatment of depression in the treatment of patients with major depressive disorder.

The safety of duloxetine and any side effects that might be associated with it.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years of age
* must be diagnosed with depression
* must sign informed consent

Exclusion Criteria:

* women who can become pregnant must be using birth control
* previous diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder
* history of substance abuse or dependence in the last year
* patients who are suicidal
* frequent or severe allergic reactions with multiple medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2003-04; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Linear measure of global benefit-risk assessment. Benefit is defined as remission at endpoint (HMAD17 total score less than or equal to 7, a virtually symptom-free state.

SECONDARY OUTCOMES:
HAMD17 Response Rates: Response is defined as a greater or equal to 50% reduction in HAMD17 total score from baseline to endpoint.
HAMD17 Time to First Response: Time to first response is defined as the visit where a sustained greater than or equal to 30% reduction in the Maier subscale of the HAMD17.
HAMD17 Remission Rates: Remission is defined as a HAMD17 total score of less than or equal to 7 at endpoint.
Hamilton Anxiety Rating Scale (HAMA) that measures the presence and severity of anxiety. The 14-item version of this scale will be used to assess the severity of anxiety and its improvement during the course of therapy.
Clinical Global Impressions of Severity (CGI-Severity) Scale to record the severity of illness at the time of assessment.
Patient's Global Impressions of Improvement (PGI Improvement) Scale is a patient-rated instrument that measures the improvement of the patient's symptoms.
HAMD17 Subscales to evaluate severity of psychic and somatic manifestations of anxiety, as well as agitation; evaluate dysfunction in mood, work, and sexual activity, as well as overall motor retardation; evaluate initial, middle and late insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta, Canada

REFERENCES:
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com